CLINICAL TRIAL: NCT02450890
Title: A Phase III, Multi-Center, Randomized, Double-blind, Placebo Controlled, Two-way Cross-over Clinical Study to Evaluate Safety and Efficacy of ORADUR®-Methylphenidate in Children and Adolescents With ADHD
Brief Title: Evaluate Safety and Efficacy of ORADUR®-Methylphenidate in Children and Adolescents With ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Orient Pharma Co., Ltd. (Industry)
Collaborators: Durect (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: OP-2PN012-301
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ORADUR®-Methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo First, then ORADUR® (Placebo Comparator): Placebo once daily for 2 weeks in Period 1 and ORADUR®-Methylphenidate oral capsule at the optimal dose once daily for 2 weeks in period 2. (No washout period between two treatment periods)
  Interventions: Drug: Placebo First, then ORADUR®
- ORADUR® First, then Placebo (Experimental): ORADUR®-Methylphenidate oral capsule at the optimal dose once daily for 2 weeks in Period 1 and Placebo once daily for 2 weeks in period 2. (No washout period between two treatment periods)
  Interventions: Drug: ORADUR® First, then Placebo

INTERVENTIONS:
Drug: Placebo First, then ORADUR® — ORADUR®-Methylphenidate is available in three dosage forms (22mg, 33mg or 44mg). The optimal dose for each subject will be determined in the open-label titration period. After randomization, subjects will be subjected to the 4-week double-blind two-way cross-over treatment phase with 2 study periods (2 weeks of placebo and 2 weeks of ORADUR®-Methylphenidate oral capsule at the optimal dose, according to a pre-determined randomization schedule).
  Other Names: Placebo
  Arms: Placebo First, then ORADUR®
Drug: ORADUR® First, then Placebo — ORADUR®-Methylphenidate is available in three dosage forms (22mg, 33mg or 44mg). The optimal dose for each subject will be determined in the open-label titration period. After randomization, subjects will be subjected to the 4-week double-blind two-way cross-over treatment phase with 2 study periods (2 weeks of placebo and 2 weeks of ORADUR®-Methylphenidate oral capsule at the optimal dose, according to a pre-determined randomization schedule).
  Other Names: Placebo
  Arms: ORADUR® First, then Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ORADUR®-Methylphenidate in children and adolescents with ADHD.

DETAILED DESCRIPTION:
This Phase III, multi-center, randomized, double-blind, placebo controlled, two-way cross-over study aims to observe the efficacy and safety of ORADUR®-Methylphenidate in children and adolescents with ADHD age 6 to 18 years old.

The study is comprised of four main phases: a screening period lasting about 14 days, an open-label titration period lasting 2 to 4 weeks, a double-blind and placebo controlled two-way cross-over study period of 4 weeks (2 weeks for Period 1 and 2 weeks for Period 2), then a follow-up phase of 2 weeks. Screening baseline is defined as Day 0 (Visit 2).

At the last day of the titration period (Day 14 for 22 mg, Day 21 for 33 mg group, and Day 28 for 44 mg group), subjects will be randomly assigned to receive ORADUR®-Methylphenidate at their optimal dose or placebo at a 1:1 ratio according to the randomization scheme during each study period (Period 1 and Period 2) at treatment phase; no washout period will be included between two treatment periods.

ELIGIBILITY:
Main inclusion criteria:

1. Female or male subjects with age between 6 and 18 years old.
2. Subjects with documented diagnosis of one of the three presentations of Attention Deficit Hyperactivity Disorder (ADHD) within one year by investigator assessment using Diagnostic & Statistical Manual for Mental Disorders-Fifth Edition (DSM-5).
3. Both subjects and parents/guardians have provided their signed and dated informed consent form for the study.

Main exclusion criteria:

1. Subjects have received ADHD treatment for over 1 year or those who have received other ADHD treatment within 30 days prior to the study treatment initiation.
2. By investigator's evaluation, subjects are very anxious, tense or agitated.
3. Subjects known to be allergic to any ORADUR®-methylphenidate ingredients.
4. Subjects with an estimated intelligence quotient (IQ) < 80.
5. Subjects are taking a concomitant medication (ex: Monoamine Oxidase Inhibitor (MAOI)) that is likely to interfere with safe administration of methylphenidate within 14 day prior to the study treatment initiation.
6. Subjects are joining other clinical studies and receiving any other investigational medical products within 30 days prior to the study treatment initiation.
7. Subjects have glaucoma (narrow angle glaucoma), on-going seizure disorder, or other psychotic disorder.
8. Subjects have chronic tics, Tourette's syndrome, or a family history of Tourette's syndrome.
9. Subjects have clinically significant gastrointestinal problems, including narrowing of the gastrointestinal tract.
10. Subjects/caregivers are (in the case of subjects whose parents/caregivers were to fill out the study questionnaires) with drug or alcohol abuse/dependence within the prior 6 months.
11. By the investigators' discretion, subjects with serious or unstable medical illness that will interfere with the evaluations of study efficacy and safety.
12. In the investigators' opinion, subjects cannot understand or follow the instructions given in the study.
13. Psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 114 (Actual)
Dates: Start 2015-06; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
SNAP-IV teacher form score in ORADUR®-Methylphenidate vs. placebo | 2 weeks
  To determine the Swanson, Nolan, and Pelham-IV (SNAP-IV) teacher form score of children and adolescents with ADHD who are administered ORADUR®-Methylphenidate versus those who are administered placebo

SECONDARY OUTCOMES:
SNAP-IV parent form score in ORADUR®-Methylphenidate (open titration period) | 2 weeks
  To examine changes of the Swanson, Nolan, and Pelham-IV (SNAP-IV) parent form scores in children and adolescents with ADHD administered ORADUR®-Methylphenidate at different dose schedules in the titration period.
SNAP-IV parent form score in ORADUR®-Methylphenidate vs. placebo | 2 weeks
  To determine the Swanson, Nolan, and Pelham-IV (SNAP-IV) parent form score of children and adolescents with ADHD who are administered ORADUR®-Methylphenidate versus those who are administered placebo.
Remission rate in ORADUR®-Methylphenidate vs. placebo | 2 weeks
  To determine the remission rate of children and adolescents with ADHD who are administered ORADUR®-Methylphenidate versus those who are administered placebo.
Conners' Teacher's Rating Scale score in ORADUR®-Methylphenidate vs. placebo | 2 weeks
  To determine the Conners' Teacher's Rating Scale score of children and adolescents with ADHD who are administered ORADUR®-Methylphenidate versus those who are administered placebo.
Conners' Continuous Performance Test (CPT-II) performance in ORADUR®-Methylphenidate vs. placebo | 2 to 4 weeks
  To determine the Conners' Continuous Performance Test (CPT-II) performance of children and adolescents with ADHD who are administered ORADUR®-Methylphenidate versus those who are administered placebo.
Diagnostic & Statistical Manual for Mental Disorders-Fifth Edition (DSM-5) diagnosis in ORADUR®-Methylphenidate vs. placebo | 2 to 4 weeks
  To determine the Diagnostic & Statistical Manual for Mental Disorders-Fifth Edition (DSM-5) diagnosis of children and adolescents with ADHD who are administered ORADUR®-Methylphenidate versus those who are administered placebo.
Clinical Global Impression-ADHD-Severity (CGI-S) score in ORADUR®-Methylphenidate vs. placebo | 2 weeks
  To determine the Clinical Global Impression-ADHD-Severity (CGI-S) score of children and adolescents with ADHD who are administered ORADUR®-Methylphenidate versus those who are administered placebo.
Clinical Global Impression-ADHD-Improvement (CGI-I) score in ORADUR®-Methylphenidate vs. placebo | 2 weeks
  To determine the Clinical Global Impression-ADHD-Improvement (CGI-I) score of children and adolescents with ADHD who are administered ORADUR®-Methylphenidate versus those who are administered placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Tai Chang, PhD, Study Director — Orient Pharma Co., Ltd.
Locations (4):
- Taiwan (4):
  - Chang Gung Medical Foundation- Chiayi Branch, Chiayi City
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Medical Foundation- Linkuo Branch, Taoyuan District

REFERENCES:
- [Derived] Shang CY, Chou TL, Hsieh CY, Gau SS. A Counting Stroop Functional Magnetic Resonance Imaging Study on the Effects of ORADUR-Methylphenidate in Drug-Naive Children with Attention-Deficit/Hyperactivity Disorder. J Child Adolesc Psychopharmacol. 2022 Nov;32(9):467-475. doi: 10.1089/cap.2022.0024. Epub 2022 Oct 14. PMID 36251766
- [Derived] Huang YS, Yeh CB, Chen CH, Shang CY, Gau SS. A Randomized, Double-Blind, Placebo-Controlled, Two-Way Crossover Clinical Trial of ORADUR-Methylphenidate for Treating Children and Adolescents with Attention-Deficit/Hyperactivity Disorder. J Child Adolesc Psychopharmacol. 2021 Apr;31(3):164-178. doi: 10.1089/cap.2020.0104. Epub 2020 Dec 31. PMID 33395356